CLINICAL TRIAL: NCT02385838
Title: Impact of Different Front-of-pack Nutrition Labels on Consumer Purchasing Intentions: Randomized Trial in the NutriNet-Santé Study
Brief Title: Impact of Nutrition Labels on Consumer Purchasing Intentions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Paris 13 (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Serge HERCBERG, Prof. Dr., University of Paris 13
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Nutrinet SM1
Record Dates: First submitted 2015-02-26; First posted 2015-03-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Food Labeling; Choice Behavior
Keywords: Nutrition labelling; Front-of-pack nutrition labels; Purchasing intentions; Nutritional quality; Randomized controlled trial (RCT)

ARMS (5):
- 5-Color Nutrition Label (5-CNL) (Experimental): The 5-CNL front-of-pack nutrition labeling is affixed on the front-of-pack of foodstuffs of the experimental web-based supermarket
  Interventions: Behavioral: 5-CNL
- Mutiple Traffic Lights (MTL) (Experimental): The MTL front-of-pack nutrition labeling is affixed on the front-of-pack of foodstuffs of the experimental web-based supermarket
  Interventions: Behavioral: MTL
- Guidelines Daily Amounts (GDA) (Experimental): The GDA front-of-pack nutrition labeling is affixed on the front-of-pack of foodstuffs of the experimental web-based supermarket
  Interventions: Behavioral: GDA
- Green Tick (Tick) (Experimental): The Tick front-of-pack nutrition labeling is affixed on the front-of-pack of foodstuffs of the experimental web-based supermarket
  Interventions: Behavioral: Tick
- No label (No Intervention): No front-of-pack nutrition labeling is affixed on the front-of-pack of foodstuffs of the experimental web-based supermarket

INTERVENTIONS:
Behavioral: 5-CNL — The 5-CNL front-of-pack nutrition label is introduced on foodstuffs in a controlled shopping environment
  Arms: 5-Color Nutrition Label (5-CNL)
Behavioral: MTL — The MTL front-of-pack nutrition label is introduced on foodstuffs in a controlled shopping environment
  Arms: Mutiple Traffic Lights (MTL)
Behavioral: GDA — The GDA front-of-pack nutrition label is introduced on foodstuffs in a controlled shopping environment
  Arms: Guidelines Daily Amounts (GDA)
Behavioral: Tick — The Tick front-of-pack nutrition label is introduced on foodstuffs in a controlled shopping environment
  Arms: Green Tick (Tick)

SUMMARY:
The purpose of this interventional study is to compare the impact of four different Front-Of-Pack (FOP) nutrition labels on purchasing intentions. This study is nested in the ongoing web-based prospective observational NutriNet-Santé cohort study, including on December 2014 around 150,000 participants. The investigators will perform a five-arm randomized trial where participants will be subjected to different FOP nutrition label formats: Guidelines Daily Amount (GDA), Multiple Traffic Lights (MTL), 5-Color Nutrition Label (5-CNL), Green Tick (Tick) and a 'no label' condition. The impact of front-of-pack nutrition labels on the nutritional quality of the shopping cart will be assessed. Participants from the NutriNet-Santé cohort study will be randomly assigned to one of these five experimental conditions according to their sociodemographic characteristics.

Purchasing intentions will be assessed using an experimental web-based supermarket designed to look like a regular online grocery store. The supermarket includes 269 unique products divided into 4 categories: dairy products, processed meat/delicatessen, savory and breakfast/sugary products. Each category is then separated into specific products families like yogurt, milk, cheese, etc. for the dairy products category. Inside a food family, the selection of foodstuffs will be made to obtain a representative sample of the products commonly sold in French supermarket. For each type of products, at least two variants are proposed. Products are retailers or manufacturers branded. Categories of products that are not usually bought each week, or which are likely to be bought from different sources are not included on the web-based supermarket.

Participants are asked to simulate a shopping situation: they have to select a week worth of food for their family among proposed products. If the user is not able to find a product he/she usually buy, the instruction is to select similar product among proposed ones.

Information provided for each product is: name, price and the picture with the FOP label/or not according to the experimental condition to which the participant is allocated. A brief explanation of the FOP label used is also given.

ELIGIBILITY:
Inclusion Criteria:

* Being a participant of the NutriNet-Santé cohort study
* Completing the preliminary questionnaire about nutrition knowledge and purchasing habits
* Completing online shopping in the experimental supermarket

Exclusion Criteria:

* Not going shopping usually
* Having a difference greater than 400€ between the price of their shopping cart versus their usual weekly shopping cart budget
* Having aberrant body mass index (i.e. >55 or <11 for women and <13 for men)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11981 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall nutritional quality of the shopping cart | up to 27 weeks
  The overall nutritional quality of the shopping cart is estimated by computing the Food Standards Agency (FSA) nutrient profiling system for 100 g of the cart (i.e. sum of the FSA score of all products, divided by the number of products chosen)

SECONDARY OUTCOMES:
Caloric value of the shopping cart | up to 27 weeks
  The caloric value of the shopping cart is calculated for 100 g of the cart
Nutrients content of the shopping cart | up to 27 weeks
  The nutrients content (i.e. lipids, saturated fatty acids, sugars, proteins, fibers, sodium) of the shopping cart is calculated for 100 g of the cart

CONTACTS AND LOCATIONS:
Overall Officials: Serge Hercberg, Pr, Principal Investigator — EREN
Locations (1):
- Equipe de Recherche en Epidémiologie Nutritionnelle, Bobigny, France

REFERENCES:
- [Derived] Ducrot P, Julia C, Mejean C, Kesse-Guyot E, Touvier M, Fezeu LK, Hercberg S, Peneau S. Impact of Different Front-of-Pack Nutrition Labels on Consumer Purchasing Intentions: A Randomized Controlled Trial. Am J Prev Med. 2016 May;50(5):627-636. doi: 10.1016/j.amepre.2015.10.020. Epub 2015 Dec 15. PMID 26699246